CLINICAL TRIAL: NCT01945320
Title: The Effects Nutrition Status and Body Composition on HD Patients' Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112008RIC
Record Dates: First submitted 2013-09-09; First posted 2013-09-18 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Body Composition; Nutritional Wasting; Malnutrition
Keywords: hemodialysis; wasting and malnutrition; nutrition status; bioelectrical impedance analysis; body composition
MeSH Terms: conditions — Malnutrition; Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HD-BCM: 1. Patients at National Taiwan University Hospital
  2. Patients who have received HD more than 3 months
  3. Patients who sign the informed consents
  4. Patients who aged between 20-90 years

SUMMARY:
A prospective long-term follow up of hemodialysis (HD) patients' outcome correlates with nutritional status and body composition. We will evaluate the body composition change among HD patients every three months with bioelectrical impedance analysis (BIA). The change of body composition will correlated with other clinical data including nutritional, inflammatory parameters and survival.

DETAILED DESCRIPTION:
Wasting and malnutrition are common and serious complications in patients on hemodialysis and are strongly associated with adverse outcomes. Techniques for assessing nutrition have limitations and, due to metabolic effects and confounding effects of altered hydration and other body composition abnormalities, these limitations are greater in the context of renal failure. Bioelectrical impedance analysis is a promising method for the objective assessment and monitoring of body composition. Body composition techniques subdivide the body into compartments on the basis of differing physical properties. The different compartments reflect hydration, nutrition/wasting, body fat, and bone mineral content, which are all of great importance in patients on hemodialysis. We will conduct a prospective long-term follow up of HD patients' outcome correlates with nutritional status and body compositions. The patients will receive BIA every three months, and other routine clinical data such as dialysis adequacy and monthly biochemical data are collected to analyze. An additional blood sample of 8 ml will be collected every 3 months during the BIA survey for other inflammatory cytokines and nutritional markers such as adiponectin, leptin, ghrelin, prealbumin, fetuin A, fructosamine, IL-1, IL-6 and transferrin. The follow up period will be as long as possible and the last recruited into this study is in the Dec. 2016. These data will be used for the morbidity and mortality analysis to see if body compositions will be more useful and timely than the other nutritional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients at National Taiwan University Hospital
* Patients who have received hemodialysis more than 3 months
* Patients who sign the informed consents

Exclusion Criteria:

* Patients who have received hemodialysis less than 3 months
* Patients who refuse to sign informed consents
* Patients who refuse to draw additional blood for research

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HD patients
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the correlation between the change of body composition by bioelectrical impedance analysis (BIA) with other clinical data including nutritional, inflammatory parameters and survival. | Participants will be tracked once every 6 months, up to 5 years to be followed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan